CLINICAL TRIAL: NCT00124553
Title: The Potential for Diet Modification to Improve Glycaemic Control and Cardiovascular Risk Factors Over and Above Drug Therapy in Type 2 Diabetes at High Risk of Cardiovascular Disease
Brief Title: LOADD (Lifestyle Over and Above Drugs in Diabetes) Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Edgar National Centre for Diabetes Research (Other)
Collaborators: University of Otago (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENCDR_1
Record Dates: First submitted 2005-07-27; First posted 2005-07-28 (Estimated); Last update posted 2007-03-28 (Estimated); Status verified 2007-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes; cardiovascular risk; glycaemic control; dietary modification
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Behavioral: Intensive dietary advice

SUMMARY:
In the past, nutritional management formed the cornerstone of treatment of type 2 diabetes (T2DM). More recently, this aspect of treatment has received less attention as drug therapy aimed not only to lower glucose, but also to treat raised blood pressure and blood fats (including cholesterol) has been more widespread. While there is evidence to suggest that blood pressure and blood fat levels have improved, overall diabetes control has not and people with diabetes appear to be becoming progressively more overweight, following trends in the general population. The proposed study involves a randomised controlled trial in which people with T2DM continuing with their regular drug treatment and surveillance, will be randomly allocated to additionally receive intensive advice regarding diet or remain on their usual treatment in this regard. The results will be judged principally in terms of body weight, waist circumference, blood pressure, blood glucose control and blood fats.

DETAILED DESCRIPTION:
This is a 6-month pilot intervention study which seeks to determine whether adherence to an intensive evidence based dietary programme, in addition to the prescription of both cardioprotective and hypoglycaemic medications recommended for patients with diabetes, will provide health benefits in terms of reducing the risk of developing or progression of complications of diabetes (particularly cardiovascular disease).

The specific aim of the project is to compare the effects of an intensive lifestyle intervention (based on the recently published evidence based recommendations of the Nutrition Study Group of the European Association for the Study of Diabetes [3]) or usual dietary advice, in diabetic patients at high risk of cardiovascular disease, treated with cardioprotective and hypoglycaemic drugs.

Study participants will be randomised into two groups:

* The control group will receive usual dietary advice and diabetes treatment from their usual GP and practice nurse (as detailed in the Management of Type 2 Diabetes and The Assessment and Management of Cardiovascular Risk guidelines published in December 2003 [1,2]).
* In addition to usual care, the intervention group will receive intensive instruction about a recommended dietary pattern based on the recently published recommendations of the Nutrition Study Group of the European Association for the Study of Diabetes [3] and where appropriate use material, for example serving size information from the above mentioned guidelines.

Outcome will be determined by examining surrogate markers of clinical endpoints. These surrogate markers will include clinical measures (weight, body mass index, blood pressure) and appropriate tests (haemoglobin A1c, fasting insulin, blood lipids, lipoproteins, inflammatory markers, and urine albumin creatinine ratio). A quality of life questionnaire will also be administered at the beginning and end of the project.

1. New Zealand Guidelines Group. The assessment and management of cardiovascular risk. Wellington, NZ. December, 2003. http://www.nzgg.org.nz
2. New Zealand Guidelines Group. Management of Type 2 diabetes. Wellington, NZ. December, 2003. http://www.nzgg.org.nz
3. Mann JI, De Leeuw I, Hermansen K, Karamanos B, Karlstrom B, Katsilambros N, Riccardi G, Rivellese AA, Rizkalla S, Slama G, Toeller M, Uusitupa M, Vessby B. Nutr Metab Cardiovasc Dis 14:373-394, 2004

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Resident in Dunedin
* Aged <70 years at the time of invitation to participate
* Most recent HbA1c level within the last 12 months ≥ 7%
* Currently prescribed oral tablets or insulin or both for glycaemic control AND three of the following: *Any pre-existing cardiovascular disease defined as a past history of myocardial infarction, angina, peripheral vascular disease, cerebrovascular accident, transient ischaemic attack; *Currently prescribed antihypertensive medication; *Currently prescribed lipid modifying medication; *Body mass index ≥25

Exclusion criteria:

* Terminal illness

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220
Dates: Start 2006-08; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Body mass index (BMI)
Glycated Haemoglobin (HbA1c)
Triglycerides
Dietary intake as measured by 3-day weighed diet records
All measures to be compared at end of study (6 months)

SECONDARY OUTCOMES:
Blood pressure
Weight
Waist circumference
Total cholesterol and lipid subfractions (LDL, HDL)
Fasting insulin
Lipoproteins A + B
Inflammatory markers
Urinary albumin:creatinine ratio
Quality of life
All measures to be compared at end of study (6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Jim I Mann, FRACP, Principal Investigator — Edgar National Centre for Diabetes Research; Kirsten Coppell, FAFPHM, Principal Investigator — Edgar National Centre for Diabetes Research
Locations (1):
- Edgar National Centre for Diabetes Research, Dunedin, Otago, New Zealand

REFERENCES:
- [Background] Mann JI, De Leeuw I, Hermansen K, Karamanos B, Karlstrom B, Katsilambros N, Riccardi G, Rivellese AA, Rizkalla S, Slama G, Toeller M, Uusitupa M, Vessby B; Diabetes and Nutrition Study Group (DNSG) of the European Association. Evidence-based nutritional approaches to the treatment and prevention of diabetes mellitus. Nutr Metab Cardiovasc Dis. 2004 Dec;14(6):373-94. doi: 10.1016/s0939-4753(04)80028-0. No abstract available. PMID 15853122
- [Background] New Zealand Guidelines Group. Assessment and Management of Cardiovascular Risk. December, 2003. Wellington, NZ. http://www.nzgg.org.nz. ISBN (print) 0-476-00091-2
- [Background] New Zealand Guidelines Group. Management of Type 2 Diabetes. Wellington, NZ. December, 2003. http://www.nzgg.org.nz. ISBN (print): 0-476-00092-0
- [Derived] Coppell KJ, Kataoka M, Williams SM, Chisholm AW, Vorgers SM, Mann JI. Nutritional intervention in patients with type 2 diabetes who are hyperglycaemic despite optimised drug treatment--Lifestyle Over and Above Drugs in Diabetes (LOADD) study: randomised controlled trial. BMJ. 2010 Jul 20;341:c3337. doi: 10.1136/bmj.c3337. PMID 20647285
- See also: Edgar National Centre for Diabetes Research website — http://www.otago.ac.nz/diabetes